CLINICAL TRIAL: NCT04618848
Title: Performance Evaluation Protocol for Sight Diagnostics' OLO CBC Analyzer by Ichilov Oncology Daily Care Center
Brief Title: Performance Evaluation Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sight Diagnostics (Industry)
Collaborators: Tel Aviv Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: PR0156
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Hematology
Keywords: Hematology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adult Oncology Patients: Adult oncology patients
  Interventions: Diagnostic Test: Fingerstick blood draw

INTERVENTIONS:
Diagnostic Test: Fingerstick blood draw — Each participant shall be pricked twice in order to perform CBC test

SUMMARY:
This study aims to establish OLO's performance accuracy of CBC results for finger prick samples across the OLO reportable range, and particularly around relevant medical decision points

DETAILED DESCRIPTION:
This study aims to establish OLO's performance accuracy of CBC results for finger prick samples across the OLO reportable range, and particularly around relevant medical decision points.

The evaluation will include two studies:

1. A matrix study will compare a capillary sample collected via finger prick with a venous sample collected into a blood tube, both scanned on OLO.
2. A method comparison study will compare Sight OLO to the site reference analyzer using a venous sample collected into a blood tube.

ELIGIBILITY:
Inclusion Criteria:

* Blood samples will be collected from oncologic patients older than 18 years old arriving at the oncologic daily care center of Ichilov hospital, with predefined normal and abnormal blood counts

Exclusion Criteria:

* Patient younger than 18 years old
* Visibly hemolyzed specimens (sample plasma should be checked for hemolysis by technician while selection of specimen from tube racks).
* Visibly clotted specimens (Reasonable to assume that samples processed with clinical reported results are not clotted).
* A sample that is not successfully scanned on OLO within 3 attempts (e.g. rejected due to irregular cell morphology, or microscopically visible hemolysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncologic patient
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
CBC Comparison | Immediately after sample collection is completed
  Comparison between CBC results obtained from the Sight OLO and the reference device in venous and capillary samples covering medical decision points relevant to onclology patient

CONTACTS AND LOCATIONS:
Overall Officials: Yochay Eshel, Principal Investigator — Sponsor GmbH

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT04618848/Prot_000.pdf